CLINICAL TRIAL: NCT03242356
Title: Oral Feeding During Established Labor. Current Practices in the Obstetric Department of the Femme Mère Enfant Hospital (Lyon, France)
Brief Title: Oral Feeding During Established Labor at Our Institution
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0454
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2017-08

CONDITIONS: Labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire to assess of the application of the current French guidelines as to fasting during labor. — Questionnaire focuses on :
  * oral intake of clear fluid during the labor
  * oral intake of solid meal during the labor
  * fasting duration for solid and liquids
  * instruction received as to fasting during labor, nature of these instructions, and who given the instruction (midwife, nurse anesthetist, …)
  * discomfort related to thirst during labor
  * discomfort related to hunger during labor
  We will also record several medical data as to the course of pregnancy and delivery, analgesia technique, history and characteristics of the parturient.

SUMMARY:
Current French guidelines allow oral intake of clear fluid in women in established labor under epidural analgesia. To date, no study assessed how these guidelines are followed in clinical practice. This study aims to assess the current practices as to the fasting during the labor at our institution, while assessing the experience and the expectations of the parturients (level of comfort or discomfort related to fasting).

ELIGIBILITY:
Inclusion Criteria:

* All adult woman who has been in labor in our hospital

Exclusion Criteria:

* Patient refusal
* Elective cesarean section, or emergency cesarean section in a woman not in labor
* Intrauterine fetal death
* Therapeutic abortion
* Patient consent not available (for example, in case of severe post-partum hemorrhage)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult women who were in labor in our hospital interviewed within 2 hours after vaginal delivery or cesarean section decided during the labor
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2017-11-25 (Actual); Study Completion 2017-11-25 (Actual)

PRIMARY OUTCOMES:
Rate of parturients who declared to have ingested clear fluid during the labor. | The survey will be completed within 2 hours following the delivery

SECONDARY OUTCOMES:
Determine the instructions given by health professionals, their spontaneous or non-spontaneous character and the information related to the given fast, according to the parturient | The survey will be completed within 2 hours following the delivery
  Determine the instructions given by health professionals, whether they are spontaneous or not
Specify the type of liquid ingested (water or sweet liquid) and its volume | The survey will be completed within 2 hours following the delivery
  Nature and volume of liquids ingested
Specify the frequency of ingestion of solid foods during labor | The survey will be completed within 2 hours following the delivery
  Nature and quantity of ingested solids
Assess the degree of discomfort associated with thirst that was felt during labor | The survey will be completed within 2 hours following the delivery
  Degree of discomfort related to thirst on a simple numeric scale (0: no discomfort at 10: very uncomfortable)
Assess the degree of discomfort associated with hunger that was felt during labor | The survey will be completed within 2 hours following the delivery
  Degree of discomfort related to hunger on a simple numeric scale (0: no discomfort at 10: very uncomfortable)
Evaluate women's satisfaction with the fasting instructions received | The survey will be completed within 2 hours following the delivery
  Satisfaction with fasting instructions given on a simple numerical scale (0: very high dissatisfaction, 10: maximum satisfaction)
Determine if nausea and vomiting are more common in women who have ingested fluids during labor | The survey will be completed within 2 hours following the delivery
  Incidence of at least one episode of nausea and vomiting during labor
Analyze the factors associated with fasting during work and their concordance with the French recommendations on fasting during labor | The survey will be completed within 2 hours following the delivery
  Analysis of independent risk factors for the patient's strict fasting during labor
Indicate the total duration of fast and solid fasting before birth | The survey will be completed within 2 hours following the delivery
  Total duration of liquid fasting and solids preceding birth
Compare fasting instructions received by patients and practices reported by professionals | The survey will be completed within 2 hours following the delivery
  Fasting instructions received by patients and practices reported by professionals obtained during a practice survey

CONTACTS AND LOCATIONS:
Locations (1):
- hopital Femme Mère Enfant, Bron, France